CLINICAL TRIAL: NCT02901366
Title: Plasma Concentration, Excretion and Mass Balance Orally Administered 14C-FYU-981 in Healthy Male Subjects
Brief Title: Mass Balance Study of FYU-981
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fuji Yakuhin Co., Ltd. (Industry)
Collaborators: Mochida Pharmaceutical Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FYU-981-009
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Healthy Male Subjects
Keywords: Mass balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14C-FYU-981 (Experimental): 14C-FYU-981, (Oral single dosing)
  Interventions: Drug: 14C-FYU-981

INTERVENTIONS:
Drug: 14C-FYU-981 — 14C-FYU-981, (Oral single dosing)

SUMMARY:
To assess the plasma pharmacokinetics, the routes extent of elimination, and the metabolites of FYU-981 after a single 1 mg oral dose of 14C-FYU-981 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy adult subjects
* Body mass index: >=18.5 and <25.0

Exclusion Criteria:

* Subjects with any disease or any history of diseases that might be unsuitable for participation in the clinical study
* Have participated in a [14C]-study within the last 12 months prior to dosing of the investigational drug
* Exposure to radiation for therapeutic or diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton) within the last 12 months prior to dosing of the investigational drug
* Occupationally exposed worker

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax: Maximum plasma concentration) | 168 hours
Pharmacokinetics (AUC: Area under the plasma concentration-time curve) | 168 hours
Pharmacokinetics (Tmax: Time to reach the peak plasma concentration) | 168 hours
Pharmacokinetics (T1/2: Elimination half-life of plasma concentration) | 168 hours
Pharmacokinetics (kel: Elimination rate constant) | 168 hours
Pharmacokinetics (Vd/F: Distribution volume / Fraction of dose absorbed | 168 hours
Pharmacokinetics (CLtot/F: Total clearance / Fraction of dose absorbed) | 168 hours
Pharmacokinetics (MRT: Mean residence time) | 168 hours
Pharmacokinetics (Ae(urine), Ae(feces) and Ae(air): Amount of radioactivity excreted in urine, feces, or air) | 168 hours or 72 hours (Ae(air))
Pharmacokinetics (fe(urine) , fe(feces) and fe(air): Fraction of radioactivity excreted in urine, feces, or air) | 168 hours or 72 hours (Ae(air))
Pharmacokinetics (Ae(total): Total amount of radioactivity excreted) | 168 hours
Pharmacokinetics (fe(total): Total fraction of radioactivity excreted) | 168 hours
Pharmacokinetics (Ae(urine + air): Amount of radioactivity excreted in urine and air) | 168 hours
Pharmacokinetics (fe(urine + air): Fraction of radioactivity excreted in urine and air) | 168 hours
Pharmacokinetics (Ratios of FYU-981 and its metabolites in plasma, urine and feces) | 168 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan